CLINICAL TRIAL: NCT04149639
Title: An Open-label Study to Investigate the Effectiveness of a LifeSeasons NeuroQ Supplement in Addition to Four Bredesen Recommended Lifestyle Changes to Improve Cognitive Function in Healthy Adults Who Have One or More Risk Factors for Cognitive Decline
Brief Title: A Study Investigating the Effectiveness of a LifeSeasons NeuroQ Supplement With Lifestyle Changes to Improve Cognitive Function in Healthy Adults Who Have One or More Risk Factors for Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeSeasons Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19IPHL
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: NeuroQ; Dr. Bredesen; PreCODE protocol; ReCODE method; cognitive decline; The End of Alzheimer's; cognitive support; cognitive health
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Open-label design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeuroQ (Experimental): Directions: take 2 capsules at the same time daily
  Interventions: Dietary Supplement: NeuroQ

INTERVENTIONS:
Dietary Supplement: NeuroQ — Supplement includes phosphatidylserine, coffee fruit, curcumin, ginkgo, gotu kola, and propolis active ingredients inside a veggie capsule.

SUMMARY:
The objective of this study is to evaluate the efficacy of a NeuroQ supplement designed by Dr. Bredesen to complement his Lifestyle modification protocol. Eligible participants will be expected to consume the NeuroQ supplement and are recommended to make lifestyle changes based on Dr. Bredesen's protocol. Forty participants are expected to enroll into the study, completing study assessments at check in visits days 30 and 60, and at the end of study visit on day 90. A brief follow up phone call will be conducted approximately 30 days after study completion to ask participants if they have continued using the lifestyle changes and if they have purchased and continued to consume the NeuroQ supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 45 years of age or older with one or more of the following risk factors for cognitive decline:

   * Self-reported genetic risk factor of Alzheimer's Disease or dementia as confirmed by Apolipoprotein 4 genetic testing
   * Self-reported family history of Alzheimer's Disease or dementia in a first-degree relative
   * Self-reported lifestyle risk factor: sedentary lifestyle; poor dietary habits (e.g. insufficient consumption of fruits and vegetables for necessary nutrients); poor social support network (e.g. majority of evenings and weekends are spent in isolation); poor stress management skills (e.g. binge eating habits or performing harmful activities during periods of stress); poor sleep habits; metabolic syndrome
   * Exception: Individuals 60 years of age or older may be enrolled without any of the above risk factors.
2. BMI between 18.5 and 32.5 kg/m2
3. Female participants are not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening

or,

Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to screening 4. Self-reported as non-smoker or user of any nicotine-containing products 5. Absence of dementia or other significant cognitive impairment as assessed by Mini Mental State Exam-2 Standard Version (MMSE-2) score ≥24 6. Participants who test between the 24-75th percentile in the in one or more domains in the NCI 7. Low frequency of depressed mood as assessed by PHQ-9 score of 4 or less 8. Agree to avoid caffeine consumption 24 hours prior to in-clinic visits 9. Agree to avoid alcohol consumption 24 hours prior to in-clinic visits 10. Healthy as determined by medical history and laboratory results as assessed by QI

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Allergy, sensitivity, or intolerance to the investigational product's (IP) active or inactive ingredients
3. Self-reported confirmation of neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation. For e.g.:

   • Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, neurodegenerative disease, infections, insomnia
4. Participants with vitamin deficiencies affecting cognition:

   * Magnesium
   * Cobalamin (Vitamin B12)
   * Folate below the normal clinical ranges, as assessed by the QI
5. Participants who test below the 24th percentile or above the 75th percentile in all domains in the NCI.
6. Current use of prescribed medications listed in Section 8.3.1.
7. Current use of over-the-counter medications, supplements, foods and/or drinks listed as concomitant medications.
8. Unstable metabolic disease or chronic diseases as assessed by the QI
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
10. Type II diabetes. Treatment on a stable dose of medication may be considered by the QI on a case by case basis
11. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case by case basis
12. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
13. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
14. Individuals who are immune-compromised
15. Verbal confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis
16. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom free for 6 months
17. Verbal confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
18. Current or history of any significant diseases of the gastrointestinal tract
19. Verbal confirmation of blood/bleeding disorders
20. Self-reported chronic use of cannabinoid products or currently taking medical cannabinoid products containing >0.3% tetrahydrocannabinol
21. Alcohol or drug abuse within the last 12 months
22. High alcohol intake (>2 drinks per day or >10 standard drinks per week)
23. Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
24. Participation in other clinical research trials 30 days prior to screening
25. Individuals who are unable to give informed consent
26. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Change in cognition as assessed by change in Neurocognitive Index (NCI) score from CNS-Vital Signs (CNS-VS) panel from screening to end-of-study. | 90-135 days
  The Neurocognitive index is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.

SECONDARY OUTCOMES:
Change in Neurocognitive Index (NCI) individual domains from screening to end-of study in participants who are fully compliant with supplementation and lifestyle modification | 90-135 days
  The Neurocognitive index is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in Neurocognitive Index (NCI) individual domains from screening to end-of-study in participants who are compliant with supplementation only | 90-135 days
  The Neurocognitive index is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in Neurocognitive Index (NCI) individual domains from screening to end-of-study in participants who are compliant with lifestyle modification only | 90-135 days
  The Neurocognitive index is an average score derived from the domain scores or a general assessment of the overall neurocognitive status of the participant. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - composite memory from screening to end-of-study | 90-135 days
  The composite memory domain measures how well subject can recognize, remember, and retrieve words and geometric figures. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - verbal memory from screening to end-of-study | 90-135 days
  The verbal memory domain measures how well subject can recognize, remember, and retrieve words. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - visual memory from screening to end-of-study | 90-135 days
  The visual memory domain measures how well subject can recognize, remember and retrieve geometric figures. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - psychomotor speed from screening to end-of-study | 90-135 days
  The psychomotor speed domain measures how well a subject perceives, attends, responds to visual-perceptual information, and performs motor speed and fine motor coordination. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - reaction time from screening to end-of-study | 90-135 days
  The reaction time domain measures how quickly the subject can react, in milliseconds, to a simple and increasingly complex direction set. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - complex attention from screening to end-of-study | 90-135 days
  The complex attention domain measures the ability to track and respond to a variety of stimuli over lengthy periods of time and/or perform mental tasks requiring vigilance quickly and accurately. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - cognitive flexibility from screening to end-of-study | 90-135 days
  The cognitive flexibility domain measures how well subject is able to adapt to rapidly changing and increasingly complex set of directions and/or to manipulate the information. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - processing speed from screening to end-of-study | 90-135 days
  The processing speed domain measures how well a subject recognizes and processes information i.e., perceiving, attending/responding to incoming information, motor speed, fine motor coordination, and visual-perceptual ability. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - executive function from screening to end-of-study | 90-135 days
  The executive function domain measures how well a subject recognizes rules, categories, and manages or navigates rapid decision making. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - simple attention from screening to end-of-study | 90-135 days
  The simple attention domain measures the participants ability to track and respond to a single defined stimulus over lengthy periods of time while performing vigilance and response inhibition quickly and accurately. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Change in individual Central Nervous System-Vital Signs (CNS-VS) domain - motor speed from screening to end-of-study | 90-135 days
  The motor speed domain measures the participants ability to perform movements to produce and satisfy an intention towards a manual action and goal. The scores range from less than 70 (very low) to above 110 (above average). A higher score means higher neurocognitive function and higher capacity.
Number of participants motivated to make lasting changes to their lifestyle at end-of-study. | 90-120 days
Change in Mini Mental State Exam Version 2 (MMSE-2) score from screening to end-of study. | 90-135 days
  The Mini Mental State Exam Version 2 is an assessment of the level of consciousness. It is a series of 30 questions scored either 0 (incorrect) or 1 (correct). The range of scores is 0 to 30. A higher value means the participant answered more questions correctly.

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events following 30-day, supplementation. | 30 days
Incidence of pre-emergent and post-emergent adverse events following 60-day, supplementation. | 60 days
Incidence of pre-emergent and post-emergent adverse events following 90-day, supplementation. | 90 days
Change in systolic blood pressure following 30-day supplementation | 30 days
Change in systolic blood pressure following 60-day supplementation | 60 days
Change in systolic blood pressure following 90-day supplementation | 90 days
Change in diastolic blood pressure following 30-day supplementation | 30 days
Change in diastolic blood pressure following 60-day supplementation | 60 days
Change in diastolic blood pressure following 90-day supplementation | 90 days
Change in heart rate following 30-day supplementation | 30 days
Change in heart rate following 60-day supplementation | 60 days
Change in heart rate following 90-day supplementation | 90 days
Change in CMP following 90-day supplementation | 90 days
Change in complete blood count following 90-day supplementation | 90 days
Change in neutrophil levels in the blood following 90-day supplementation | 90 days
  Units: XE9/L
Change in lymphocyte blood levels following 90-day supplementation | 90 days
  Units: XE9/L
Change in monocyte blood levels following 90-day supplementation | 90 days
  Units: XE9/L
Change in eosinophil blood levels following 90-day supplementation | 90 days
  Units: XE9/L
Change in basophil blood levels following 90-day supplementation | 90 days
  Units: XE9/L
Change in red blood cell (RBC) count following 90-day supplementation | 90 days
Change in hemoglobin levels in the blood following 90-day supplementation | 90 days
  Units: g/L
Change in hematocrit levels in the blood following 90-day supplementation | 90 days
  Units: L/L
Change in platelet count following 90-day supplementation | 90 days
Change in mean corpuscular volume (MCV) following 90-day supplementation | 90 days
Change in mean corpuscular hemoglobin (MCH) following 90-day supplementation | 90 days
  Units: pg
Change in mean corpuscular hemoglobin concentration (MCHC) following 90-day supplementation | 90 days
Change in red cell distribution width (RDW) following 90-day supplementation | 90 days
Difference in brain activity as measured by quantitative electroencephalography (qEEG) from baseline to end-of-study in 10 participants. | 90 days
  Alpha, Beta, Delta, and Theta bandwidths will be analyzed using the eVox system.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Langston, Study Director — LifeSeasons Inc.
Locations (2):
- United States (2):
  - Kapoor Medical Center, Studio City, California
  - LifeSeasons Medical Center, Flower Mound, Texas

IPD SHARING:
Plan to Share IPD: No